CLINICAL TRIAL: NCT06953466
Title: A Single Center, Open Label, Expanded Access Study of QRX003 Lotion in Subjects With Netherton Syndrome
Brief Title: Clinical Study of QRX003 Lotion in Subjects With Netherton Syndrome
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Quoin Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-QRX003-003; Sponsor Funded (Other: Quoin Pharmaceuticals, Ltd.)
Record Dates: First submitted 2025-04-07; First posted 2025-05-01 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Netherton Syndrome
MeSH Terms: conditions — Netherton Syndrome

STUDY DESIGN:
Intervention Model Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- QRX003, 4% BID (Experimental): Subjects will apply test article twice daily (BID) for 12 weeks
  Interventions: Drug: QRX003, 4% Lotion

INTERVENTIONS:
Drug: QRX003, 4% Lotion — QRX003 Topical Lotion containing 4% active drug (serine protease inhibitor)

SUMMARY:
The goal of this clinical trial (via an expanded access Treatment Protocol) is to learn if QRX003 (an investigational drug) applied topically to the skin (including up to the entire body [except the scalp]) works to treat the genetic disease Netherton syndrome. It will also learn about the safety of QRX003. The main questions the trial aims to answer are:

1. Does QRX003 impact the clinical presentation of NS in adults and minors by improving the clinical symptoms (diseased skin area, itch, and discomfort; based on clinical scoring, subject self-assessment, and other criteria)?
2. What medical problems do participants have when taking QRX003?
3. What percent of subjects will require rescue therapy?

Participants will:

Take drug QRX003 twice daily (applied topically to all affected areas of the body excluding the scalp) for 3 months, visit the clinic once every 4-6 weeks for checkups and tests, and to keep a dosing diary that records the times they applied the drug.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or non-pregnant female at least 14 years of age.
2. Females must be post-menopausal , surgically sterile , or use an effective method of birth control , for the duration of the study and for 3 months following completion of treatment. Women of childbearing potential (WOCBP) must have a negative urine pregnancy test (UPT) at Visit 1/Screening and Visit 2/Baseline.
3. Subject has a clinical diagnosis of NS and agrees to genetic testing at Visit 1/Screening for confirmation of NS diagnosis if the subject does not have test results confirming a SPINK5 mutation.
4. Subject is in good general health and free of any disease state or physical condition that might impair evaluation of NS or exposes the subject to an unacceptable risk by study participation.
5. Subject is on a stable treatment regimen including topical therapy for NS prior to baseline that is expected to remain stable for the duration of the study

Exclusion Criteria:

1. Subject is pregnant, lactating, or is planning to become pregnant during the study.
2. Subject has any skin pathology in the Treatment Area or condition that, could interfere with the evaluation of the test article or requires use of interfering topical, systemic, or surgical therapy.
3. Subject has active cancer of any type excluding non-melanoma skin cancer outside of the Treatment Area.
4. Subject has diabetes of any type, except non-insulin dependent diabetes mellitus that is reasonably controlled.
5. Subject has evidence of active infection during screening, or serious infection within 30 days prior to Visit 2/Baseline.
6. Subject has known human immunodeficiency virus, hepatitis B or C virus, or active or latent tuberculosis.
7. Subject has used ultraviolet phototherapy within the Treatment Area within 10 weeks prior to Visit 2/Baseline.
8. Subject has used topical prescription treatment in the Treatment Area within 10 weeks prior to Visit 2/Baseline.
9. Subject has used any topical steroid prescription treatments in the Treatment Area within 10 weeks prior to Visit 2/Baseline.
10. Subject is currently enrolled in an investigational drug, biologic, or device study.
11. Subject has used an investigational drug, biologic, or device treatment within 30 days prior to Visit 2/Baseline.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with 1-point reduction on IGA | Up to week 16
  Description: Proportion of subjects with 1-point reduction on the Investigator's Global Assessment (IGA) from Baseline. The IGA assesses overall severity of a subject's NS based on a 5-point scale where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe.

OTHER OUTCOMES:
Proportion of subjects with 2-point reduction on IGA | Up to week 16
  Proportion of subjects with 2-point reduction in IGA from Baseline.
NS surface area change | Up to week 16
  Change from Baseline in total Body Surface Area (BSA) affected by NS in the Treatment Area
WI-NRS score change | Up to week 16
  Change from Baseline in the Worst Itch-Numeric Rating Scale (WI-NRS) score ≥4. Itch severity is graded on an 11-point scale where 0 represents "no itch" and 10 represents "worst itch imaginable".
Safety Assessment-AEs | Up to week 16
  Any local and systemic AEs (Adverse Events)/serious AEs

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided